CLINICAL TRIAL: NCT02926859
Title: Enhancing Recovery in Early Schizophrenia - a Multi-center, Two-arm, Double-blind, Randomized Phase II Trial Investigating Cannabidiol vs. Placebo as an add-on to an Individualized Antipsychotic Treatment
Brief Title: Enhancing Recovery in Early Schizophrenia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBD-ESPRIT
Record Dates: First submitted 2016-07-07; First posted 2016-10-06 (Estimated); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (Experimental): Cannabidiol as add-on to individualized pharmacological treatment
  Interventions: Drug: Cannabidiol as add-on
- Placebo (Placebo Comparator): Placebo as add-on to individualized pharmacological treatment
  Interventions: Drug: Placebo as add-on

INTERVENTIONS:
Drug: Cannabidiol as add-on — Cannabidiol capsules 2x200 mg twice a day as add-on to individualized pharmacological treatment with either amisulpride, aripiprazole, olanzapine, quetiapine or risperidone over 26 weeks
  Arms: Cannabidiol
Drug: Placebo as add-on — Placebo capsules 2x200 mg twice a day as add-on to individualized pharmacological treatment with either amisulpride, aripiprazole, olanzapine, quetiapine or risperidone over 26 weeks
  Arms: Placebo

SUMMARY:
Current antipsychotic treatments of schizophrenia are only partially effective, and their use is often associated with serious side effects. Cannabidiol is a natural counterpart of the psychoactive component of marijuana, delta-9- tetrahydrocannabinol and has no psychotomimetic or addictive properties. In a controlled clinical trial of cannabidiol versus amisulpride in acute paranoid schizophrenia we showed a statistically significant clinical improvement in all symptoms clusters of schizophrenia compared to baseline with either treatment. Cannabidiol displayed a significantly superior side-effect profile in particular regarding prolactin elevation, extrapyramidal symptoms and weight gain. The favorable side-effect profile and potentially novel mechanism of action identify this molecule as a potential antipsychotic. However, long-term safety and efficacy data is still lacking. This study is to evaluate the efficacy and safety of the novel compound cannabidiol in the maintenance treatment of schizophrenia in comparison to placebo as an add-on to an established treatment with either amisulpride, aripiprazole, olanzapine, quetiapine or risperidone, in a 12-months, double-blind, parallel-group, randomized, placebo-controlled clinical trial. Thereby, relevant data on cannabidiol's antipsychotic potential will be gained.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent given by the subject
* DSM-IV-TR diagnosis of schizophrenic psychosis (295.10-30, 295.90)
* First documented diagnosis of schizophrenia must not be no older than seven years.
* Patients must receive a stable dose of amisulpride, aripiprazole, olanzapine, quetiapine or risperidone (TAU: treatment as usual) at least 4 weeks prior to inclusion in the study to ensure that the maximal effect of the previous medication has been received.
* Initial PANSS total score of ≤ 75 at baseline.
* proper contraception in female patients of childbearing potential
* body mass index between 18 and 40.

Exclusion Criteria:

* Lack of accountability
* positive urine drug-screening for illicit drugs at screening (except cannabinoids and benzodiazepines)
* serious suicidal risk at screening visit
* other relevant interferences of axis 1 according to diagnostic evaluation (MINI) including residual forms of schizophrenia.
* other relevant neurological or other medical disorders
* pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-04-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
All-cause discontinuation | within 12 month

SECONDARY OUTCOMES:
Improvement in Psychopathology assessed by PANSS | 6, 9 and 12 month
  Positive and Negative Syndrome Scale (PANSS)
Improvement in Psychopathology assessed by CGI | 6, 9 and 12 month
  Clinical Global Impression (CGI)
Improvement in Psychopathology assessed by BSI-53 | 6, 9 and 12 month
  Brief Symptom Inventory (BSI-53)
Improvement in Psychopathology assessed by FROGS | 6, 9 and 12 month
  Functional Remission of General Schizophrenia (FROGS)
Changes from baseline in Depression Scale | 6, 9 and 12 month
  Calgary Depression Scale for Schizophrenia (CDSS)
Improvement in social and occupational functioning assessed by GAF | 6, 9 and 12 month
  Global Assessment of Functioning (GAF)
Improvement in social and occupational functioning assessed by PSP | 6, 9 and 12 month
  Personal and Social Performance Scale (PSP)
Improvement in social and occupational functioning assessed by EMA | 6, 9 and 12 month
  Ecological Momentary Assessment (EMA)
Improvement in Quality of life assessed by WHOQUOL-Bref | 6, 9 and 12 month
  WHO Quality of Life-Bref (WHOQUOL-Bref)
Improvement in Quality of life assessed by LQLP | 6, 9 and 12 month
  Lancashire Quality of Life Profile (LQLP)
Changes from baseline in Neurocognition assessed by B-CATS | 6, 9 and 12 month
  Brief Cognitive Assessment Tool for Schizophrenia (B-CATS)
Changes from baseline in Neurocognition assessed by BACS | 6, 9 and 12 month
  Brief Assessment of Cognition in Schizophrenia (BACS)
Changes from baseline in Neurocognition assessed by UPSA-B | 6, 9 and 12 month
  University of California San Diego Performance based Skills Assessment (UPSA-B)
Changes from baseline in Neurocognition assessed by MASC | 6, 9 and 12 month
  Movie for the Assessment of Social Cognition (MASC)
Changes from baseline in Neurocognition assessed by PFA | 6, 9 and 12 month
  Pictures of Facial Affect (PFA)
Treatment adherence | 6, 9 and 12 month
Changes in Cumulative dose of concomitant or rescue medication | 6, 9 and 12 month
Changes of Biomarker: alterations of endocannabinoids and lipdomic profiling | 6, 9 and 12 month

OTHER OUTCOMES:
Side effects: weight gain | 6, 9 and 12 month
  Body Mass Index, abdominal girth
Side effects: Vital Signs | 6, 9 and 12 month
  heart rate, blood pressure, electrocardiography
Side effects: UKU Side Effect rating scale | 6, 9 and 12 month
Side effects: Abnormal Involuntary Movement Scale (AIMS) | 6, 9 and 12 month
Side effects: Evaluation of extrapyramidal symptoms (EPS) | 6, 9 and 12 month
Side effects: physical and neurological examination | 6, 9 and 12 month
Standard blood tests | 6, 9 and 12 month
Columbia Suicidality Sverity Rating Scale (C-SSRS) | 6, 9 and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: F. Markus Leweke, MD, Principal Investigator — Central Institute of Mental Health
Locations (6):
- Germany (6):
  - Dep. of Psychiatry and Psychotherapy, Central Institute of Mental Health, Mannheim, Baden-Wurttemberg
  - Dept. of Psychiatry and Psychotherapy, Ludwig-Maximillians-University Munich, Munich, Bavaria
  - Dept. of Psychiatry and Psychotherapy, Charité, Campus Charité-Mitte, Berlin, B
  - Department of Psychiatry, Psychotherapy, and Psychosomatics, RWTH Aachen, Aachen, North Rhine-Westphalia
  - Dept. of Psychiatry and Psychotherapy, University Hospital of Cologne, Cologne, North Rhine-Westphalia
  - Department of Psychiatry und Psychotherapy, University Hospital Hamburg-Eppendorf, Hamburg